CLINICAL TRIAL: NCT00001927
Title: Study of Abnormal Acquired and Genetic Coagulation Factors in Children With Porencephaly and Stroke
Brief Title: Study of Abnormal Blood Clotting in Children With Stroke
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990045; 99-N-0045
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-04

CONDITIONS: Abnormalities; Blood Coagulation Disorder; Brain Disease; Cerebrovascular Accident; Vascular Disease
Keywords: Factor V Leiden; Prothrombin Mutation; Antiphospholipids; Cerebral Infarction; Thrombophilia; Porencephaly; Perinatal Stroke; Healthy Mothers; Healthy Children
MeSH Terms: conditions — Congenital Abnormalities; Blood Coagulation Disorders; Brain Diseases; Stroke; Vascular Diseases; Cerebral Infarction; Thrombophilia; Porencephaly

SUMMARY:
Effective treatment and prevention strategies for childhood stroke and porencephaly can only be developed once the causes are understood. There is increasing evidence that inherited and acquired coagulation abnormalities alone or in combination with environmental factors, predispose to arterial and venous thrombosis. Inherited abnormalities of factor V Leiden, prothrombin, protein C, protein S, and antithrombin III may account for many of these thromboses. At present there is little information on the existing distribution of these coagulation anomalies in children with thrombosis. Recent reports also suggest that these clotting abnormalities may be responsible for some instances of intracranial hemorrhage, porencephaly, cerebral palsy and fetal death.

This study will measure the frequency of several coagulation factor abnormalities (factor V Leiden, prothrombin 20210A, protein C, protein S, antithrombin III, and antiphospholipid antibodies) in children with a history of porencephaly and stroke, and will compare these to the prevalence of these mutations in population controls and family members. We will also describe the exogenous conditions which in concert with these coagulation factors, may have led to the development of thrombosis in these children....

DETAILED DESCRIPTION:
OBJECTIVES:

Effective treatment and prevention strategies for childhood stroke and porencephaly can only be developed once the causes are understood. There is increasing evidence that inherited and acquired coagulation abnormalities, alone or in combination with environmental factors, predispose to arterial and venous thrombosis. Inherited abnormalities of factor V leiden, prothrombin, protein C, protein S, and antithrombin III may account for many of these thromboses. At present there is little information on the existing distribution of these coagulation anomalies in children with thrombosis. Recent reports suggest that these clotting abnormalities may be responsible for some instances of intracranial hemorrhage, porencephaly, cerebral palsy and fetal death.

The objectives of this protocol are: 1) to determine the frequency of coagulation abnormalities in children with porencephaly or stroke as compared to healthy children, 2) to determine the frequency of coagulation abnormalities in children with porencephaly or stroke as compared to their family members, 3) to determine the frequency of coagulation abnormalities in mothers of children with stroke as compared to mothers of healthy children, and 4) to describe the exogenous conditions, which in concert with coagulation factors, may have led to the development of thrombosis in children with stroke.

STUDY POPULATION:

This study will examine: 1) children with a history of porencephaly or stroke, 2) their biological mothers, fathers, and siblings, 3) healthy volunteer children, and 4) healthy volunteer mothers.

DESIGN:

This is a case-control study conducted at the National Institute of Neurological Disorders and Stroke. Children with a history of porencephaly or stroke before 18 years of life, their first-degree relatives, healthy volunteer children, and healthy volunteer mothers will be enrolled. Each subject may complete a blood draw, buccal smear, questionnaire, and/or review of medical records depending on their study group.

OUTCOME MEASURES:

This study will measure the frequency of several coagulation factors among the study's different population groups as well as examine the exogenous conditions that may have contributed to stroke in these children. Analysis will be descriptive and quantitative.

ELIGIBILITY:
* INCLUSION CRITERIA:

CHILDREN WITH A HISTORY OF PORENCEPHALY OR STROKE:

1. Children less than 18 years of age with a history of porencephaly or cerebral infarction (stroke).
2. Children less than 18 years of age with a history of spastic hemiplegic or quadriplegic cerebral palsy (ICD-9 codes 343.1, 343.2, 343.3, 343.4, 343.8 and 343.9) with radiographic evidence of porencephaly or stroke.
3. A diagnosis of porencephaly as defined by a fluid-filled cavity within the cerebral hemispheres which may or may not communicate with CSF spaces and confirmed by at least one imaging method including computed tomography (CT), magnetic resonance (MR) and or Doppler ultrasonography.
4. A diagnosis of cerebral infarction (stroke) as defined by a new focal neurologic deficit lasting greater than or equal to 24 hours and presumably due to a vascular process (ICD-9 codes 430-437) and confirmed by brain imaging, either computed tomography (CT), magnetic resonance (MR) or Doppler ultrasonography.
5. Informed consent of the parent.
6. Informed assent of the child, when available.

FIRST-DEGREE RELATIVES OF CHILDREN WITH PORENCEPHALY OR STROKE:

1. Full biological first-degree relatives of children with a history of porencephaly or stroke enrolled in this study.
2. Informed consent of each participant.
3. Informed assent of each participant under 18 years, when available.

HEALTHY CHILDREN:

1. Children less than 18 years of age.
2. Informed consent of the parent.
3. Informed assent of the child when available.

HEALTHY MOTHERS:

1. Women between 18 and 45 years of age.
2. History of full-term pregnancy.
3. Informed consent of the participant.

EXCLUSION CRITERIA:

CHILDREN WITH A HISTORY OF PORENCEPHALY OR STROKE:

1. Children greater than 18 years of age.
2. Maternal history of cocaine abuse during pregnancy.
3. History of cancer.
4. History of other chromosomal or metabolic disorder.
5. History of trauma and or child abuse.
6. Isolated subdural hematomas.
7. History of aneurysm or vascular malformations.
8. Congenital heart disease.
9. Sickle cell disease.
10. History of CNS infection.

HEALTHY CHILDREN:

1. Children greater than 18 years of age.
2. Maternal history of cocaine abuse during pregnancy.
3. History of cancer.
4. History of other chromosomal or metabolic disorder.
5. History of trauma and or child abuse.
6. Isolated subdural hematomas.
7. History of aneurysm or vascular malformations.
8. Congenital heart disease.
9. Sickle cell disease.
10. History of CNS infection.
11. History of stroke or porencephaly.

HEALTHY MOTHERS:

1. Volunteer has biological children without a history of cancer, head trauma, aneurysm, chromosomal or metabolic disorder, congenital heart disease, sickle cell disease, meningitis or encephalitis, or stroke.
2. Cocaine use during pregnancy.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 1999-02-22; Study Completion 2011-05-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Griffin JH, Evatt B, Zimmerman TS, Kleiss AJ, Wideman C. Deficiency of protein C in congenital thrombotic disease. J Clin Invest. 1981 Nov;68(5):1370-3. doi: 10.1172/jci110385. PMID 6895379
- [Background] Allaart CF, Poort SR, Rosendaal FR, Reitsma PH, Bertina RM, Briet E. Increased risk of venous thrombosis in carriers of hereditary protein C deficiency defect. Lancet. 1993 Jan 16;341(8838):134-8. doi: 10.1016/0140-6736(93)90003-y. PMID 8093743
- [Background] Poort SR, Rosendaal FR, Reitsma PH, Bertina RM. A common genetic variation in the 3'-untranslated region of the prothrombin gene is associated with elevated plasma prothrombin levels and an increase in venous thrombosis. Blood. 1996 Nov 15;88(10):3698-703. PMID 8916933